CLINICAL TRIAL: NCT00373360
Title: Rapid Switch From Intravenous Epoprostenol to Intravenous Remodulin® (Treprostinil Sodium) in Patients With Stable Pulmonary Arterial Hypertension: Safety, Efficacy and Treatment Satisfaction
Brief Title: Safety, Efficacy and Treatment Satisfaction in Patients With PAH Rapidly Switched From Epoprostenol to Remodulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIV-PH-411
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Results first posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2013-01

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; PAH; Remodulin; treprostinil; Quality of Life; Rapid Switch
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil; Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: treprostinil sodium

INTERVENTIONS:
Drug: treprostinil sodium — rapid switch from intravenous epoprostinol to intravenous remodulin on the CADD ambulatory pump
  Other Names: Remodulin; Flolan

SUMMARY:
The purpose of this 8-week study is to compare the effects of switching from therapy with epoprostenol or Flolan to IV Remodulin. This study will also assess the effect that changing to Remodulin will have on patient satisfaction with their treatment and impact on quality of life.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH), which is defined as an elevation in pulmonary arterial pressure and pulmonary vascular resistance, is a severe hemodynamic abnormality common to a variety of diseases and syndromes. Elevation in pulmonary arterial pressure causes an increase in right ventricular afterload, impairing right ventricular function and ultimately leading to inactivity and death. The goal of PAH treatment is to lengthen survival time, to ameliorate symptoms of PAH and to improve health related quality of life (HRQOL).

Remodulin® (treprostinil sodium), a stable analogue of prostacyclin, possesses potent pulmonary and systemic vasodilatory and platelet anti-aggregatory actions in vitro and in vivo. Recently, Remodulin received FDA approval for intravenous therapy based upon bioequivalence of the IV and SC routes of administration. Remodulin is more chemically stable than epoprostenol and may offer potential safety and convenience advantages compared to intravenous epoprostenol that may impact Health Related Quality of Life (HRQOL) and/or patient satisfaction. Unlike epoprostenol, Remodulin does not need to be mixed daily and is stable at room temperature eliminating the need for ice packs. Furthermore, since Remodulin remains in the body longer than epoprostenol (4 hrs instead of less than 5 minutes) there is less risk of cardiovascular collapse from a sudden interruption of infusion, such as a line clog. In an open-label study in Europe, patients who were using a type of portable medication pump called the CADD Legacy pump were rapidly switched from Flolan to Remodulin with no serious side effects. This study will examine effects of switching from therapy with epoprostenol or Flolan to IV Remodulin and compare changes in HRQOL and treatment satisfaction before and after rapid switch from epoprostenol to Remodulin in patients with pulmonary hypertension using the CADD legacy pump.

Participation in this study will last approximately 10 weeks. Study procedures include routine blood tests, medical history, physical exams, disease evaluation, exercise tests and patient questionnaires. Participants will have 4 visits during the study and will spend at least 1 night in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 70 years
* Diagnosis of Idiopathic or Familial Pulmonary Arterial Hypertension (PAH)or PAH associated with a collagen vascular disease or PAH associated with congenital systemic-to-pulmonary shunt repaired greater than 5 years prior to study entry or PAH associated with portal hypertension with mild or moderate hepatic dysfunction (Grade of A or B on the Child-Pugh Classification Scale)or PAH associated with drug or toxins or CTEPH
* WHO Class II-III
* Currently receiving intravenous epoprostenol therapy for at least three months and a stable dose for at least one month.
* Have central intravenous catheter
* Optimally treated with conventional pulmonary hypertension therapy and clinically stable for at least one month.
* Mentally and physically capable of learning to administer Remodulin using an intravenous infusion pump.

Exclusion Criteria:

* Nursing or pregnant woman
* Have any other type of PAH due to conditions other than noted in the above inclusion criteria, including but not limited to PAH related to thrombotic or embolic disease
* Have any other disease that is associated with pulmonary hypertension (e.g. sickle cell anemia, schistosomiasis)
* Changes to chronic PAH therapy (i.e., new therapy added within last 30 days[including but not limited to oxygen, a different category of vasodilator, a diuretic, digoxin, bosentan, sildenafil] or PAH medication discontinued within 7 days of study entry.
* Received any prostacyclin or prostacyclin analog except epoprostenol in the past 3 months.
* Central venous line infection within the past 30 days.
* Previous documented evidence of significant parenchymal lung disease
* Evidence or history of left-sided heart disease
* Musculoskeletal disorder or any other disease, which is thought to limit ambulation, or be connected to a machine that is not portable
* Uncontrolled hypertension, chronic renal insufficiency, or active infection.
* Use of investigational drug within past 30 days.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omar Minai, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject participated in this study between July 2007 and January 2008.
Pre-assignment Details: All subjects were required to be receiving continuous intravenous epoprostenol therapy for at least three months and at a stable dose for at least thirty days prior to enrollment in this study.
Groups:
- Treprostinil Sodium: All subjects received active treatment with treprostinil sodium.
Period: Overall Study
Arm/Group | Treprostinil Sodium
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
PAH Etiology [Number; unit: participants]
  Idiopathic PAH | 7
  Connective Tissue Disease (CTD) | 2
  Other | 1
World Health Organization (WHO) Functional Classification for PAH [Number; unit: participants] — Class I: No limitation of physical activity. Class II: Slight limitation of physical activity. Class III: Marked limitation of physical activity. Class IV: Inability to carry out any physical activity without symptoms.
  participants
    Class II | 6
    Class III | 4
Six minute walk distance [Mean (Full Range); unit: meters] | 447.7 [195 to 663]
Epoprostenol dose [Mean (Full Range); unit: ng/kg/min] | 27.15 [15 to 58]

OUTCOME MEASURES:

1. Primary Outcome: Change in the Distance Transversed During the 6 Minute Walk Test From Baseline to Week 8.
Time Frame: Baseline and Week 8
Population: As this was a small open label study, the statistics applied to the results were descriptive. For all efficacy endpoints, data obtained from study assessments during the treatment phase were compared to Baseline.
  assessments
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
meters | -2.2 (34.8)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 1.000, Wilcoxon signed rank test

2. Secondary Outcome: Change in Borg Dyspnea Score Immediately After Six Minute Walk Test From Baseline to Week 8
Description: The Borg dyspnea score is a 10-point scale rating the maximum level of dyspnea experienced during the 6-minute walk test. The Borg dyspnea score was assessed immediately following the 6-minute walk test. Scores ranged from 0 (for no shortness of breath) to 10 (for greatest shortness of breath ever experienced).
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
units on a scale | 1.56 (0.98)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.008, Wilcoxon signed rank test

3. Secondary Outcome: Change in World Health Organization (WHO) Functional Classification of PAH From Baseline to Week 8
Description: Class I: Patients with pulmonary hypertension but without resulting limitation of physical activity. Ordinary physical activity does not cause undue dyspnea or fatigue, chest pain, or near syncope.
  Class II: Patients with pulmonary hypertension resulting in slight limitation of physical activity. These patients are comfortable at rest, but ordinary physical activity causes undue dyspnea or fatigue, chest pain or near syncope.
  Class III: Patients with pulmonary hypertension resulting in marked limitation of physical activity. They are comfortable at rest. Ordinary activity causes undue dyspnea or fatigue, chest pain, or near syncope.
  Class IV: Patients with pulmonary hypertension with inability to carry out any physical activity without symptoms. These patients manifest signs of right heart failure. Dyspnea and/or fatigue may be present even at rest. Discomfort is increased by any physical activity.
Time Frame: Baseline and Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 11
  No Change | 89
  Worsened | 0
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 1.000, Wilcoxon signed rank test

4. Secondary Outcome: Change in Symptoms of Dyspnea From Baseline to Week 8
Description: The presence or absence of dyspnea was documented. If present, the intensity of dyspnea was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 22
  No Change | 33
  Worsened | 44
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.531, Wilcoxon signed rank test

5. Secondary Outcome: Change in Symptoms of Edema From Baseline to Week 8
Description: The presence or absence of edema was documented. If present, the intensity of edema was rated mild, moderate, or severe.
Time Frame: Baseline to Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 22
  No Change | 56
  Worsened | 22
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 1.000, Wilcoxon signed rank test

6. Secondary Outcome: Change in Symptoms of Orthopnea From Baseline to Week 8
Description: The presence or absence of orthopnea was documented. If present, the intensity of orthopnea was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 22
  No Change | 78
  Worsened | 0
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.500, Wilcoxon signed rank test

7. Secondary Outcome: Change in Symptoms of Dizziness From Baseline to Week 8
Description: The presence or absence of dizziness was documented. If present, the intensity of dizziness was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 11
  No Change | 89
  Worsened | 0
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 1.000, Wilcoxon signed rank test

8. Secondary Outcome: Change in Symptoms of Fatigue From Baseline to Week 8
Description: The presence or absence of fatigue was documented. If present, the intensity of fatigue was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 22
  No Change | 67
  Worsened | 11
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change from Baseline to Week 8; Test type: Superiority or Other; p = 1.000, Wilcoxon signed rank test

9. Secondary Outcome: Change in Symptoms of Syncope From Baseline to Week 8
Description: The presence or absence of syncope was documented. If present, the intensity of syncope was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 0
  No Change | 100
  Worsened | 0
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0, Wilcoxon signed rank test

10. Secondary Outcome: Change in Symptoms of Chest Pain From Baseline to Week 8
Description: The presence or absence of chest pain was documented. If present, the intensity of chest pain was rated mild, moderate, or severe.
Time Frame: Baseline and Week 8
Measure: Number; unit: percentage of participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
percentage of participants
  Improved | 0
  No Change | 89
  Worsened | 11
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 1.000, Wilcoxon signed rank test

11. Secondary Outcome: Change in Effectiveness Score on Treatment Satisfaction Scale From Baseline to Week 8
Description: The Treatment Satisfaction Questionnaire for Medication (TSQM) is a validated instrument that measures four major dimensions of patient satisfaction with medications: effectiveness, side effects, convenience, and global satisfaction. TSQM Scale scores are computed by adding the items loading on each factor. The lowest possible score is subtracted from this composite score and divided by the greatest possible score minus the lowest possible score. This provided a transformed score between 0 and 1 that should be multiplied by 100 (scale 0-100). A low score indicates low satisfaction and a high score indicates high satisfaction with treatment.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
units on a scale
  Effectiveness Score at Baseline | 71.6 (29.2)
  Effectiveness Score at Week 8 | 82.7 (23.1)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.031, Wilcoxon signed rank test

12. Secondary Outcome: Change in Side-Effects Score on Treatment Satisfaction Scale From Baseline to Week 8
Description: as for outcome 11
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
units on a scale
  Side Effects Score at Baseline | 71.5 (14.4)
  Side Effects Score at Week 8 | 84.7 (12.1)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.031, Wilcoxon signed rank test

13. Secondary Outcome: Change in Convenience Score on Treatment Satisfaction Scale From Baseline to Week 8
Description: as for outcome 11
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
units on a scale
  Convenience Score at Baseline | 59.9 (14.4)
  Convenience Score at Week 8 | 90.7 (10.8)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.004, Wilcoxon signed rank test

14. Secondary Outcome: Change in Global Satisfaction Score on Treatment Satisfaction Scale From Baseline to Week 8
Description: as for outcome 11
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
units on a scale
  Global Satisfaction Score at Baseline | 84.1 (15.1)
  Global Satisfaction Score at Week 8 | 92.1 (14.0)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.063, Wilcoxon signed rank test

15. Secondary Outcome: Change in Total Score on Quality of Life Questionnaire From Baseline to Week 8
Description: The Cambridge Pulmonary Hypertension Outcome Review (CAMPHOR) is a health related quality of life instrument specific to PAH. The total score can range from 0 -75; the higher the score, the worse the outcome.
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
units on a scale
  CAMPHOR score at Baseline | 18.9 (12.5)
  CAMPHOR score at Week 8 | 12.9 (10.8)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change Between Baseline and Week 8; Test type: Superiority or Other; p = 0.203, Wilcoxon signed rank test

16. Secondary Outcome: Change in Patient Impression of Change in Symptoms of PAH From Baseline to Week 8
Description: Subjects were asked to compare their symptoms of PAH as compared to 8 weeks prior and rate as much better, somewhat better, about the same, somewhat worse, or much worse.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
participants
  Much better | 5
  Somewhat better | 1
  About the same | 3
  Somewhat worse | 0
  Much worse | 0

17. Secondary Outcome: Change in Patient Impression of Change on Time Spent Dealing With Therapy From Baseline to Week 8
Description: Subjects were asked to compare their previous experience with Flolan and rate how much time was spent dealing with intravenous Remodulin therapy as much less, somewhat less, about the same, somewhat more, or much more.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
participants
  Much less | 8
  Somewhat Less | 0
  About the same | 1
  Somewhat more | 0
  Much more | 0

18. Secondary Outcome: Change in Patient Impression of Change of Satisfaction With Therapy From Baseline to Week 8
Description: Subjects were asked to compare their previous experience with Flolan and rate satisfaction with intravenous Remodulin therapy over the past two weeks as much more satisfied, more satisfied, about the same, less satisfied, or much less satisfied.
Time Frame: Baseline and Week 8
Measure: Number; unit: participants
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
participants
  Much more satisfied | 7
  More satisfied | 2
  About the same | 0
  Less satisfied | 0
  Much less satisfied | 0

19. Secondary Outcome: Change in Total Weekly Time Spent to Gather/Set-up Materials Associated With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
minutes
  Time to gather/set up epoprostenol at Baseline | 34.9 (28.7)
  Time to gather/set up Remodulin at Week 8 | 27.0 (28.7)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change from Baseline to Week 8; Test type: Superiority or Other; p = 0.250, Wilcoxon signed rank test

20. Secondary Outcome: Change in Total Weekly Time Spent to Connect Drug With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
minutes
  Time spent to connect epoprostenol at Baseline | 23.2 (14.4)
  Time spent to connect Remodulin at Week 8 | 18.7 (13.9)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.207, Wilcoxon signed rank test

21. Secondary Outcome: Change in Total Weekly Time Spent to Change Dressing With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
minutes
  Time to change dressing with epoprostenol at BL | 31.4 (14.2)
  Time to change dressing with Remdoluin at Wk 8 | 28.6 (25.8)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.297, Wilcoxon signed rank test

22. Secondary Outcome: Change in Total Weekly Time Spent to Prepare Drug With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
minutes
  Time to prepare epoprostenol at Baseline | 109.0 (61.0)
  Time to prepare Remodulin at Week 8 | 47.8 (31.6)
Statistical Analysis 1: Comparison: Treprostinil Sodium; Change between Baseline and Week 8; Test type: Superiority or Other; p = 0.004, Wilcoxon signed rank test

23. Secondary Outcome: Change in Total Number of Times Daily Required to Disconnect Infusion Pump With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: number of times per day
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
number of times per day
  Disconnect pump at Baseline (epoprostenol) | 7.7 (5.3)
  Disconnect pump at Wk 8 (Remodulin) | 4.1 (1.9)

24. Secondary Outcome: Change in Total Number of Times Daily Required to Check Infusion Pump With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: number of times per day
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
number of times per day
  Check pump at Baseline (epoprostenol) | 19.2 (11.5)
  Check pump at Week 8 (Remodulin) | 12.2 (8.9)

25. Secondary Outcome: Change in Total Number of Times Daily Infusion Pump Alarms With Intravenous Remodulin Therapy Compared to Same Activities With Intravenous Epoprostenol
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: number of times per day
Arm/Group | Treprostinil Sodium
Number analyzed (Participants) | 9
number of times per day
  Daily alarms at Baseline (epoprostenol) | 2.4 (3.3)
  Daily alarms at Week 8 (Remodulin) | 0.8 (1.1)

ADVERSE EVENTS:
Arm/Group | Treprostinil Sodium
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Sodium (N=10)
Gastroenteritis (Gastrointestinal disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treprostinil Sodium (N=10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Headache (General disorders) | 2 (2)
Restless Leg Syndrome (Nervous system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hand fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Injection site erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Peripheral edema (Vascular disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
catheter site inflammation (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days